CLINICAL TRIAL: NCT06407245
Title: Efficacy of Exercise Snacks in Real-World Settings in Individuals Living With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-03417
Record Dates: First submitted 2024-04-19; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Snacks (Experimental): Vigorous-intensity bodyweight exercises performed 4 times per day on at least 5 days per week.
  Interventions: Other: Exercise Snacks
- Placebo Exercise (Active Comparator): Low-intensity stretching exercises performed 4 times per day on at least 5 days per week.
  Interventions: Other: Placebo Exercise

INTERVENTIONS:
Other: Exercise Snacks — The "movement breaks" will be individualized to exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues) and adaptable to multiple environments (e.g., home, work) delivered via mobile phone application.
  Arms: Exercise Snacks
Other: Placebo Exercise — The "movement breaks" will be individualized to exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues) and adaptable to multiple environments (e.g., home, work) delivered via mobile phone application.
  Arms: Placebo Exercise

SUMMARY:
To conduct a pilot randomized control trial to determine the feasibility of a 12-week, technology-enabled exercise snacks intervention in adults living with type 2 diabetes in a real-world setting. We will also assess preliminary efficacy based on measures of glycemic control and fitness.

DETAILED DESCRIPTION:
Participants will be randomized into an Exercise Snacks or a Placebo Exercise group for 12 weeks. The former will involve bodyweight exercises performed with vigorous effort and the latter will involve low-intensity exercises. Following baseline testing, individualized interventions will be delivered at home or work via customized mobile application ("app") or web platform. Participants will be instructed to perform a minimum of 4 isolated bouts of prescribed exercises per day on at least 5 days per week. Each bout will be one minute in duration. The interventions will be individualized and consider exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues), and be adaptable to multiple environments (e.g., home, work). To facilitate this, participants will have a pre-intervention meeting wherein any physical limitations will be documented, and a research assistant will discuss the prescribed intervention and determine when and where the participants will plan to perform their exercises. After 12 weeks, participants will be asked to return to the lab for follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-75 years.
2. Have physician-diagnosed type 2 diabetes.
3. Physically inactive (performing <150 min moderate-to-vigorous physical activity per week).
4. Body mass index: 18.5-40 kg/m2.
5. Taking ≤3 glucose-lowering medications (excluding insulin) and stable dose for > 6 months.
6. Taking ≤2 commonly prescribed cardiovascular medications (e.g., statins, antihypertensive).
7. HbA1c ≤8.5%.
8. Able to maintain current physical activity patterns during the study.
9. Cleared to engage in physical activity using the Get Active Questionnaire and, if applicable, consultation with a health care provider or Qualified Exercise Professional.
10. Access to a computer, tablet or smartphone for intervention delivery and tracking.
11. Ability to read and write in English.

Exclusion Criteria:

1. Chronic musculoskeletal condition or recent (within 2 years) cardiovascular event preventing participation in exercise.
2. Lack of internet access.
3. Angina upon exertion assessed by the Rose Angina Questionnaire.
4. Prescribed beta-blockers that can compromise the validity of heart rate measurements. during the submaximal exercise test.
5. Have uncontrolled high blood pressure (hypertension; ≥ 160/90 mmHg) or an atypical blood pressure or pulse rate at rest or during exercise as determined by a physician.
6. Have a scheduled surgical procedure within the next 3-4 months that would prevent exercise participation.
7. Currently diagnosed with a cardiac or pulmonary disease (e.g., angina, arrythmia, exercise-induced bronchospasm) that would prevent exercise participation.
8. Have a psychiatric disorder that could prevent you from completing the study procedures or visits.
9. Have donated more than 0.5 L of blood within the last 4 weeks.
10. Currently following an extreme diet (e.g., very low carbohydrate/calorie, ketogenic) or taking dietary/nutritional supplements that impact glucose control (e.g., exogenous ketones).
11. Currently have diabetic ulcers, peripheral vascular disease, or diabetic neuropathy that will prevent participation in exercise.
12. Currently participating in another clinical trial that interferes with the study procedures.
13. Currently on dialysis.
14. Currently pregnant or planning on becoming pregnant during the intervention (i.e., within the next 4 months).
15. Have had an episode of severe hypoglycemia in the past 6 months (defined as having neurological symptoms consistent with neuroglycopenia and required assistance in treatment by a second party).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
Determine the number of individuals living with type 2 diabetes that are eligible to participate in the trial | NA (recruitment period)
  The number of participants approached and reasons for not joining the study.
Determine the number of eligible individuals who would be willing to take part in this trial | NA (recruitment period)
  The number of patients who enrol.
Determine the number and percentage of participants retained after the 12-week intervention | after the 12-week intervention
  Number and percentage of patients who drop-out and reasons.
Determine the number of one-minute exercise bouts performed during the 12-week intervention | during the 12 weeks
  Number of exercise bouts performed each week of the intervention.

SECONDARY OUTCOMES:
Change in glycated hemoglobin measured before and after the 12-week intervention | 0-12 weeks
  Glycated hemoglobin (A1c) at baseline and after 12 weeks.
Change in fasting glucose measured before and after the 12-week intervention | 0-12 weeks
  Fasting glucose measured at baseline and after the 12-week intervention.
Change in fasting insulin measured before and after the 12-week intervention | 0-12 weeks
  Fasting insulin measured at baseline and after the 12-week intervention
Change in 24h glucose concentration | before (week 0; before the intervention) and week 11 of the intervention
  Average of 24h glucose value measured with continuous glucose monitor at week 0 and week 11 of the intervention.
Change in cardiorespiratory fitness measured before and after the 12-week intervention | 0-12 weeks
  Submaximal YMCA cycle ergometer test to estimate VO2 peak.
Change in lower body muscular endurance measured before and after the 12-week intervention | 0-12 weeks
  The 30-second sit-to-stand pre- and post-intervention.
Change in upper body maximal strength measured before and after the 12-week intervention | 0-12 weeks
  Grip strength test using a hand dynamometer pre- and post-intervention
Change in body composition measured before and after the 12-week intervention | 0-12 weeks
  Waist circumference, weight and body mass index assessed pre- and post- intervention.
Change in blood pressure measured before and after the 12-week intervention | 0-12 weeks
  Seated systolic and diastolic blood pressure measured before and after the 12-week intervention.
Change in blood lipid profile measured before and after the 12-week intervention | 0-12 weeks
  Total cholesterol, high-density lipoprotein (HDL) cholesterol, Non-HDL cholesterol, low-density lipoprotein (LDL) cholesterol, and Triglycerides.
Change in complete blood count measured before and after the 12-week intervention | 0-12 weeks
  Red blood cells, white blood cells, haemoglobin, haematocrit, and platelet.
Change in plasma inflammatory cytokines measured before and after the 12-week intervention | 0-12 weeks
  TNF-α, IL-6, IL-10, CRP
Change in health-related quality of life measured before and after the 12-week intervention | 0-12 weeks
  Euro Quality of Life 5 Dimension 5 Level (EQ-5D-5L) questionnaire pre- and post-intervention
Changes in diabetes distress measured before and after the intervention 12-week intervention | 0-12 weeks
  Diabetes Distress Scale (DDS) questionnaire pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No